CLINICAL TRIAL: NCT06954064
Title: Digital Phenotyping of Emotional Resilience Factors to Stress in Adolescents and Young Adults: a Longitudinal Ecological Approach
Brief Title: The Student Living Lab: Intensive Longitudinal ESM Study for DP of ERFs to Stress in AYAs
Status: Enrolling by invitation | Type: Observational
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor PhD, Babes-Bolyai University
Other Study IDs: REThinkRESILIENT-DP
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Emotional Resilience

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and young adults: Adolescents and young adults will be recruited from various schools and university programs in Cluj-Napoca.
  Interventions: Other: No intervention will be applied.

INTERVENTIONS:
Other: No intervention will be applied. — No intervention will be implemented in this study, as the questionnaires will serve an exploratory purpose.

SUMMARY:
This study aims at collecting continuous mobile-based devices data for determining emotional resilience factors and childhood abuse load profiles for stress and mental health problems.

DETAILED DESCRIPTION:
Participants included in this study (age range = 10-24, G*power estimated N = 255) will complete a set of questionnaires on constructs related to mental health and resilience, creating a digital phenotype based on individual profiles and investigating the dynamics between variables over a months' period.

ELIGIBILITY:
Inclusion Criteria:

* adolescents and young adults between 10 and 24 years old provided with written parental consent where applicable

Exclusion Criteria:

* intellectual disability or physical limitations precluded the use of the computer program

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: School- and university-aged students recruited from educational institutions in Cluj-Napoca.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Resilience factors | One month, weekly (5 administrations)
  The Rugged Resilience Measure (RRM) is a 10-item scale measuring internal essential qualities associated with resilience, using 5-point Likert scales for scoring, from 1 = not at all to 5 = a lot.
Mental Health | One month, weekly (5 administrations)
  The Depression, Anxiety, and Stress Scales (DASS-21) are comprised of 21 items measuring the frequency of symptoms that can be bothering individuals in the sphere of depression, anxiety and stress. The scoring is based on Likert scales from 0 = Never to 4 = Almost always.

CONTACTS AND LOCATIONS:
Overall Officials: Oana A. David, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No